CLINICAL TRIAL: NCT03203265
Title: Thai Red Cross AIDS Research Centre (TRCARC)
Brief Title: Innovative Strategy to Offer Online Test and Treat for Thai MSM/TG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: amfAR GMT Implementation Research Grant (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: amfAR Test and Treat
Record Dates: First submitted 2017-05-25; First posted 2017-06-29 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2019-10

CONDITIONS: HIV/AIDS
Keywords: HIV home testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective study to evaluate the first-time HIV testing, successful referral to HIV treatment, retention HIV testing among 3 different study groups. A participants will receive offline HIV testing,counseling and conventional retention strategies. HIV-positive result in A can choose to have either online or offline to HIV treatment. B1 participants will be guided to access services at the 'Adam's Love Clinic, that set up specifically to provide private, fast HIV testing and post-test counseling. B2 participants will be mailed a rapid HIV test kit. Counselor will guide the participant through an online HIV testing process. Post-test counseling will provided HIV test result online. Participants can choose one of two HIV testing and post-test counseling options. HIV-positive participants in B1 and B2 can choose again to refer to HIV treatment either online or offline. All participants in B1 and B2 will receive an online retention strategy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A:Offline HIV testing and counseling (Other): Participants in Group A will be invited to come to the Thai Red Cross Anonymous Clinic, RSAT or SWING drop-in centers in Bangkok, or SWING or Sisters drop-in centers in Pattaya. After registration, they will receive standard HIV Testing and Counseling (HTC) services.
  Interventions: Other: Group A: Offline HTC
- B1:Offline (Other): participants will be guided to access services at the 'Adam's Love Offline Clinic,' a clinic set up specifically to provide private and fast HIV testing and post-test counseling only.
  Interventions: Other: Group B1: Offline HIV testing and post-test counseling
- B2: Online (Other): participants will be mailed a rapid HIV test kit. A trained online counselor will guide the participant through an online HIV testing process which includes quality checking of the test kit, obtaining blood through finger prick, performing the testing steps, and reading the test result.
  Interventions: Other: Group B2: Online HIV testing and post-test counseling

INTERVENTIONS:
Other: Group A: Offline HTC — Offline or online referral to HIV treatment facility HIV-positive participants can choose to receive either an offline or online referral to HIV treatment facilities. An offline referral method usually includes a referral letter and/or a telephone call, followed by a series of calls to participants to ensure successful referral. Those who choose an online referral will be able to register online with an HIV treatment facility which provides ART without cost under the national programs. Participants will receive a registration code which will allow them to access HIV treatment clinics directly without the need to go through the regular registration and appointment system at that facility.
  Arms: A:Offline HIV testing and counseling
Other: Group B1: Offline HIV testing and post-test counseling — participants will be guided to access services at the 'Adam's Love Offline Clinic,' a clinic set up specifically to provide private and fast HIV testing and post-test counseling only referred from the Adam's Love Online Clinic.
  Arms: B1:Offline
Other: Group B2: Online HIV testing and post-test counseling — A trained online counselor will guide the participant through an online HIV testing process which includes quality checking of the test kit,obtaining blood through finger prick,performing the testing steps,reading the test result. A positive result from the first test will trigger the need for referral to confirmatory tests. The provisional nature of the positive result from the single rapid HIV test will be emphasized but the urgency to get immediate confirmatory tests and linkage to HIV treatment facilities will encouraged and supported. HIV positive test result will be confirmed only with three positive tests. Any online testing session with uncertain qualities at any step will be repeated at a later time or the participant will be offered offline HIV testing.
  Arms: B2: Online

SUMMARY:
This study will ask Thai MSM and transgender women (TG) participants to self-select to participate in one of the 3 different study groups which provide various degrees of integrated online interventions and offline interventions for the Recruit-Test-Treat-Retain for HIV prevention and care among 3 groups (A, B1 and B2). All participants will be followed up either offline or online for 12 months. HIV-negative participants will be scheduled for repeat HTC at months 6 and 12. HIV-positive participants will be scheduled either offline or online to review their treatment history at months 6 and 12. HIV-negative participants in Group B1 and B2 can choose again at months 6 and 12 to switch from the online to offline, and vice versa, at the HIV testing/post-test counseling step and the referral to HIV treatment step

ELIGIBILITY:
Inclusion Criteria:

1. Thai national
2. Age >18 years
3. Men or transgender women who have at least 1 unprotected anal sex with men within the past 6 months
4. Live in the Bangkok Metropolitan Region (Bangkok, Pathumthani, Samutprakarn, Samutsakorn, Nakornpathom and Nonthaburi) or Pattaya
5. Not known to be HIV-positive, i.e., never tested for HIV or previous HIV test(s) negative
6. Willing to participate in the study for 12 months.
7. Provide verbal informed consent

Exclusion Criteria:

1. Known HIV-positive serostatus

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-04-06 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
The proportion of first-time HIV testers, proportion of successful HIV tests completed, proportion of successful referral to HIV treatment, and retention rate. | 1 Years
  The first-time HIV testers, successful HIV tests completed and successful referral to HIV treatment are the categorical data which don't have the units to measure. These variables are the binary outcome in which there are only two possible status e.g. yes or no, therapeutic successes or failure. The details are as follows:
  * The first-time HIV testers: this outcome variable is collected from the questionnaire; the probability of the outcome is likely to be "yes" or "no".
  * Successful HIV tests completed: this outcome variable is collected form the result of the laboratory; the probability of the outcome is likely to be "complete" or "incomplete".
  * Successful referral to HIV treatment: this outcome variable is collected form the confirmation of antiretroviral treatment; the probability of the outcome is likely to be "successful" or "failure".
  Therefore frequency and proportions of participants who have the possible outcome that we are interested (who are the first HIV testers, who

SECONDARY OUTCOMES:
The proportion of HIV-positive participants who have virological suppression at each study visit after initiating ART. | 1 Years
  The proportion of HIV-positive participants who have virological suppression at each study visit after initiating ART among MSM and TG who access online vs. offline services will be reported together with 95% confidence intervals. Formal comparisons between groups will be made using a Chi-squared test.
The retention rates of HIV-negative MSM and TG for repeated HIV testing and HIV-positive MSM and TG for antiretroviral treatment when online vs. offline retention methods are used | 1 Years
  The retention rate (or event-free survival functions) is the probability value that participant will remain in the study in any time point. The probability value is between 0 to 100% and will be estimated using Kaplan-Meier method for overall and separately by HIV-status and arms. Formal comparisons between HIV-status, online and offline retention arms will be made by a log-rank test.
The factors associated with the preferences for the online option of HIV pre-test counseling, HIV testing and post-test counseling, referral for HIV treatment, and retention services among MSM and TG | 1 Years
  The association of covariates with a preference for online vs. offline services at first visit will be modeled using logistic regression. Predictor covariates will include socio-demographic data, sexual and drug use behaviors, social network characteristics, perceived barriers and facilitators for HIV testing, beliefs and experiences around stigma and discrimination related to HIV and/or being MSM or TG, strengths and supports for stigma/discrimination, and HIV testing history.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre (TRCARC)
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Derived] Phanuphak N, Jantarapakde J, Himmad L, Sungsing T, Meksena R, Phomthong S, Phoseeta P, Tongmuang S, Mingkwanrungruang P, Meekrua D, Sukthongsa S, Hongwiangchan S, Upanun N, Jirajariyavej S, Jadwattanakul T, Barisri S, Pankam T, Phanuphak P. Linkages to HIV confirmatory testing and antiretroviral therapy after online, supervised, HIV self-testing among Thai men who have sex with men and transgender women. J Int AIDS Soc. 2020 Jan;23(1):e25448. doi: 10.1002/jia2.25448. PMID 31960589
- [Derived] Phanuphak N, Anand T, Jantarapakde J, Nitpolprasert C, Himmad K, Sungsing T, Trachunthong D, Phomthong S, Phoseeta P, Tongmuang S, Mingkwanrungruang P, Meekrua D, Sukthongsa S, Hongwiangchan S, Upanun N, Barisri J, Pankam T, Phanuphak P. What would you choose: Online or Offline or Mixed services? Feasibility of online HIV counselling and testing among Thai men who have sex with men and transgender women and factors associated with service uptake. J Int AIDS Soc. 2018 Jul;21 Suppl 5(Suppl Suppl 5):e25118. doi: 10.1002/jia2.25118. PMID 30033644